CLINICAL TRIAL: NCT06562179
Title: A Prospective, Single-Center Investigation of the da Vinci SP® Surgical System in Hepatopancreaticobiliary and Foregut Operations for Benign and Malignant Disease.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Principal Investigator, Sharona B. Ross, MD, MD, Foregut and HPB Surgeon, AdventHealth
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1907766
Record Dates: First submitted 2024-07-29; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Hepatopancreaticobiliary and Foregut Operations
Keywords: SP DaVinci; Gallbladder removal; Esophageal procedures; Gastric resections; Pancreas procedures; Liver procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- da Vinci SP® Single-Port Robotic Surgical System (Experimental): This study will be separated into four stages, depending on the condition the participant is diagnosed with. Each Participant will go through (1) one operation.
  Stage One will include five (5) subjects who undergo cholecystectomy and five (5) subjects who undergo hiatal hernia repair with fundoplication (Nissen or Toupet) for a total of ten (10) subjects.
  Stage Two will include five (5) subjects who undergo gastrectomy and five (5) subjects who undergo distal pancreatectomy for a total of ten (10) subjects.
  Stage Three will include five (5) subjects who undergo pancreaticoduodenectomy and five (5) subjects who undergo esophagectomy for a total of ten (10) subjects.
  Stage Four will include five (5) subjects who undergo hepatectomy
  Interventions: Device: da Vinci SP® Single-Port Robotic Surgical System

INTERVENTIONS:
Device: da Vinci SP® Single-Port Robotic Surgical System — The da Vinci SP® Surgical System is designed to enable the performance of surgical procedures using a minimally invasive single-port approach. The system consists of a Surgeon Console, a Vision Cart, and a Patient Cart and is used with a camera, instruments, and accessories.

SUMMARY:
The purpose of this study is to collect data to evaluate safety and performance of the da Vinci SP Surgical System, Instruments and Accessories in hepatopancreatic biliary (HPB) and Foregut operations. HPB and Foregut operations of this study consist of cholecystectomy, fundoplication, gastrectomy, distal pancreatectomy, pancreaticoduodenectomy, esophagectomy, and hepatectomy.

ELIGIBILITY:
Inclusion Criteria

Cholecystectomy Stage 1 - Inclusion Criteria:

* Patients between the ages of 18 and 80 years of age
* Either male or female
* BMI ≤ 26 kg/m2
* ASA ≤ 3
* Diagnosed with benign disease

Fundoplication Stage 1- Inclusion Criteria:

* Patients diagnosed with GERD and/or hiatal hernia
* Patients between the ages of 18 and 80 years of age
* Either men or women
* BMI ≤ 26 kg/m2
* ASA ≤ 3

Gastrectomy Stage 2- Inclusion Criteria:

* Patients between the ages of 18 and 80 years of age
* Either men or women
* BMI ≤ 26 kg/m2
* ASA ≤ 3
* Diagnosed with benign or relatively early malignant disease of the stomach
* AJCC 8th edition T0 or T1 tumor pathology
* AJCC 8th edition T2, T3, tumor pathology (following neoadjuvant therapy if necessary) at the discretion of the investigator
* Free of metastatic disease

Distal Pancreatectomy Stage 2- Inclusion Criteria:

* Patients between the ages of 18 and 80 years of age
* Either men or women
* BMI ≤ 26 kg/m2
* ASA ≤ 3
* Diagnosed with benign or malignant disease of the pancreas
* No vascular involvement
* Free of metastatic disease

Pancreaticoduodenectomy Stage 3- Inclusion Criteria:

* Patients between the ages of 18 and 80 years of age
* Either men or women
* BMI ≤ 26 kg/m2
* ASA ≤ 3
* Diagnosed with benign or malignant disease of the pancreas
* Diagnosed with benign or malignant distal bile duct disease
* No vasculature involvement (i.e., no T4 disease, pancreatic or Stage 4a or b disease, or distal bile duct Stage 3b or 4 disease)
* Free of metastatic disease

Esophagectomy Stage 3- Inclusion Criteria:

* Patients between the ages of 18 and 80 years of age
* Either men or women
* BMI ≤ 26 kg/m2
* ASA ≤ 3
* Diagnosed with benign or malignant disease of the esophagus
* AJCC 8th edition T0, T1a, T1b, T2 (without other indications for neoadjuvant therapy) tumor pathology
* AJCC 8th edition some T2, T3, or T4a, (following neoadjuvant therapy) at the discretion of the investigator
* Free of metastatic disease

Hepatectomy Stage 4- Inclusion Criteria:

* Patients between the ages of 18 and 80 years of age
* Either men or women
* BMI ≤ 26 kg/m2
* ASA ≤ 3
* Diagnosed with benign or malignant disease of the liver or bile duct
* Free of metastatic disease, not including metastatic disease to the liver (e.g., colorectal liver metastases)

Exclusion Criteria

Cholecystectomy Stage 1- Exclusion Criteria:

* Subject requiring an emergent operation
* Pregnancy or nursing
* BMI > 26 kg/m2
* Previous abdominal surgery
* Subjects with malignant disease
* Inability to provide informed consent
* Contraindicated for general anesthesia or minimally invasive surgery

Fundoplication Stage 1- Exclusion Criteria:

* Subject requiring an emergent operation
* Pregnancy or nursing
* BMI > 26 kg/m2
* Previous abdominal surgery
* Inability to provide informed consent
* Contraindicated for general anesthesia or minimally invasive surgery

Gastrectomy Stage 2- Exclusion Criteria:

* Subject requiring an emergency operation
* Pregnancy or nursing
* BMI > 26 kg/m2
* Previous abdominal surgery
* Inability to provide informed consent
* Contraindicated for general anesthesia or minimally invasive surgery
* AJCC 8th edition T2, T3, T4a, T4b tumor pathology (without neoadjuvant therapy unless contraindicated)
* Clinical or radiological evidence of distant metastatic disease

Distal Pancreatectomy Stage 2- Exclusion Criteria:

* Subject requiring an emergent operation
* Pregnancy or nursing
* BMI > 26 kg/m2
* Previous abdominal surgery
* Inability to provide informed consent
* Contraindicated for general anesthesia or minimally invasive surgery
* Tumor involvement with surrounding vasculature (e.g., common hepatic artery, superior mesenteric artery, superior mesenteric vein, portal vein)
* Clinical or radiological evidence of metastatic disease

Pancreaticoduodenectomy Stage 3- Exclusion Criteria:

* Subject requiring an emergent operation
* Pregnancy or nursing
* BMI > 26 kg/m2
* Previous abdominal surgery
* Inability to provide informed consent
* Contraindicated for general anesthesia or minimally invasive surgery
* Tumor involvement with surrounding vasculature (e.g., T4a for pancreatic disease: common hepatic artery, superior mesenteric artery, superior mesenteric vein, portal vein)
* Tumor involvement with surrounding vasculature (e.g., T3b for bile duct disease: common hepatic artery, superior mesenteric artery, superior mesenteric vein, portal vein)
* Clinical or radiological evidence of metastatic disease

Esophagectomy Stage 3- Exclusion Criteria:

* Subject requiring an emergency operation
* Pregnancy or nursing
* BMI > 26 kg/m2
* Previous abdominal surgery
* Inability to provide informed consent
* Contraindicated for general anesthesia or minimally invasive surgery
* AJCC 8th edition T2 (in some circumstances), T3, and T4a tumor pathology (without neoadjuvant therapy)
* Clinical or radiological evidence of distant metastatic disease

Hepatectomy Stage 4- Exclusion Criteria:

* Subject requiring an emergency operation
* Pregnancy or nursing
* BMI > 26 kg/m2
* Previous abdominal surgery
* Inability to provide informed consent
* Contraindicated for general anesthesia or minimally invasive surgery
* Perihilar cholangiocarcinoma (i.e., Klatskin tumor)
* Involvement of major vasculature (ex: portal vein, hepatic artery, or inferior vena cava)
* Clinical or radiological evidence of metastatic disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Completion Using the planned da Vinci SP-assisted Single Port Robot. | 12 months
  The number of subjects who completed the planned da Vinci SP-assisted operation without conversion to an alternate approach. Conversion to an alternate approach comprises conversion to open, multiport laparoscopic, multiport robotic or hand-assisted approach requiring undocking of the da Vinci SP Surgical System in order to complete the planned operation using the alternate approach.
Intraoperative and post-operative adverse events | 24 months
  The incidence of all intraoperative and post-operative adverse events that occur through the 24-month follow-up period.
Number of Positive resection Margins | 24 months
  Number of positive resection margins in patients with Malignant disease.
Number of Lymph node yield | 24 Months
  Number of lymph node yield in patients with Malignant disease.

SECONDARY OUTCOMES:
Physical Status Classification | Pre-Operative Visit
  Assessment of the fitness of patient before surgery using the ASA Physical Status Score:
  Class I - A patient in normal health Class II - A patient with mild systemic disease resulting in no functional limitations Class III - A patient with severe systemic disease that limits activity, but is not incapacitating Class IV - A patient with severe systemic disease that is a constant threat to life Class V - A moribund patient not likely to survive without the operation Class VI - A patient already declared brain dead whose organs are being removed for donor purposes
Charlson Comorbidity Index Score | Pre-Operative Visit
  Predicts one-year mortality for patients with a range of comorbid conditions, helping the physician determine how aggressively to treat a condition.
  This index score is assessed by assigning points (1,2,3 or 6) based on the likelihood of dying associated to 17 different conditions (co-morbidities). Scores are summed to provide a total score to predict mortality. Comorbidity classification is categorized as low (score ≤ 3), moderate (score 4 and 5), high (score 6 and 7), and very high comorbidity (score ≥ 8)
Operative Time | Intraoperative
  Measured in minutes
Estimated blood loss | Intraoperatively
  Measured after surgery in milliliters of blood. Estimated based on blood infusion volume during the surgery.
Intraoperative complications | Intraoperatively
  Incidence rate - number of intraoperatively complications during surgery.
Postoperative complications | 10 day, 2 months post surgery
  Incidence number of complications, assessed through electronic medical records (EMR) at 10 days 60 days post-surgery.
Post surgery complications | 2 months post surgery
  Rate of complications collected in the electronic medical using the Clavien-Dindo classification system for grading adverse events.
  Classification of surgical complications:
  Grade I - Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions.
  Grade II - Requiring pharmacological treatment with drugs. Blood transfusions and total parenteral nutrition are also included
  Grade III - Requiring surgical, endoscopic or radiological intervention Grade IIIa - Intervention not under general anesthesia Grade IIIb - Intervention under general anesthesia
  Grade IV - Life threatening complication (including Central Nervous System (CNS) complications) requiring IC/ICU management Grade IVa - Single organ dysfunction (including dialysis) Grade IVb - Multiorgan dysfunction
  Grade V - Death of a patient
In-hospital mortality | 10 days post-surgery
  Has patient expired during in-hospital stay post-surgery.
Date of Discharge | 10 days post-surgery
  Measured in number of days
Survival | 10 days, 2, months, annually through year 5
  Assessed through follow-up visits. Data collected through patient's chart in the electronic medical record (EMR).
Disease reoccurrence | 10 day, 2 month and annually through year 5
  Review of EMR records for new diagnosis assessed at schedule visits. Measured in number of days until reoccurrence diagnosis is noted in the patients' record.
30-Day Readmission | 30 days post surgery
  Review of EMR records for any readmission following discharge post surgery
30-day complications | 30 days post surgery
  Assessed as number of complications experienced by patient in the 30-day period post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Sharona Ross, MD, Principal Investigator — AdventHealth
Locations (1):
- AdventhHealth, Tampa, Florida, United States

REFERENCES:
- [Result] Rosemurgy A, Wilfong C, Craigg D, Co F, Sucandy I, Ross S. The Evolving Landscape of Esophageal Cancer: A Four-Decade Analysis. Am Surg. 2019 Sep 1;85(9):944-948. PMID 31638504
- [Result] Golkar FC, Ross SB, Sperry S, Vice M, Luberice K, Donn N, Morton C, Hernandez JM, Rosemurgy AS. Patients' perceptions of laparoendoscopic single-site surgery: the cosmetic effect. Am J Surg. 2012 Nov;204(5):751-61. doi: 10.1016/j.amjsurg.2011.07.026. PMID 23140831
- [Result] Ross S, Rosemurgy A, Albrink M, Choung E, Dapri G, Gallagher S, Hernandez J, Horgan S, Kelley W, Kia M, Marks J, Martinez J, Mintz Y, Oleynikov D, Pryor A, Rattner D, Rivas H, Roberts K, Rubach E, Schwaitzberg S, Swanstrom L, Sweeney J, Wilson E, Zemon H, Zundel N. Consensus statement of the consortium for LESS cholecystectomy. Surg Endosc. 2012 Oct;26(10):2711-6. doi: 10.1007/s00464-012-2478-y. Epub 2012 Aug 31. PMID 22936433
- [Result] Ross S, Roddenbery A, Luberice K, Paul H, Farrior T, Vice M, Patel K, Rosemurgy A. Laparoendoscopic single site (LESS) vs. conventional laparoscopic fundoplication for GERD: is there a difference? Surg Endosc. 2013 Feb;27(2):538-47. doi: 10.1007/s00464-012-2476-0. Epub 2012 Jul 18. PMID 22806533
- [Result] Sukharamwala P, Teta A, Ross S, Co F, Alvarez-Calderon G, Luberice K, Rosemurgy A. Over 250 Laparoendoscopic Single Site (LESS) Fundoplications: Lessons Learned. Am Surg. 2015 Sep;81(9):870-5. PMID 26350663
- [Result] Rosemurgy AS, Downs D, Swaid F, Ross SB. Laparoendoscopic Single-Site (LESS) Nissen Fundoplication: How We Do It. J Gastrointest Surg. 2016 Dec;20(12):2093-2099. doi: 10.1007/s11605-016-3290-0. Epub 2016 Oct 11. No abstract available. PMID 27730403
- [Result] Ryan CE, Ross SB, Sukharamwala PB, Sadowitz BD, Wood TW, Rosemurgy AS. Distal pancreatectomy and splenectomy: a robotic or LESS approach. JSLS. 2015 Jan-Mar;19(1):e2014.00246. doi: 10.4293/JSLS.2014.00246. PMID 25848192
- [Result] Barbaros U, Sumer A, Demirel T, Karakullukcu N, Batman B, Icscan Y, Saricam G, Serin K, Loh WL, Dinccag A, Mercan S. Single incision laparoscopic pancreas resection for pancreatic metastasis of renal cell carcinoma. JSLS. 2010 Oct-Dec;14(4):566-70. doi: 10.4293/108680810X12924466008448. PMID 21605524
- [Result] Rosemurgy AS, Ross SB, Espeut A, Nguyen D, Crespo K, Syblis C, Vasanthakumar P, Sucandy I. Survival and Robotic Approach for Pancreaticoduodenectomy: A Propensity Score-Match Study. J Am Coll Surg. 2022 Apr 1;234(4):677-684. doi: 10.1097/XCS.0000000000000137. PMID 35290288
- [Result] Rosemurgy A, Ross S, Bourdeau T, Craigg D, Spence J, Alvior J, Sucandy I. Robotic Pancreaticoduodenectomy Is the Future: Here and Now. J Am Coll Surg. 2019 Apr;228(4):613-624. doi: 10.1016/j.jamcollsurg.2018.12.040. Epub 2019 Jan 23. PMID 30682410
- [Result] Rosemurgy A, Ross S, Bourdeau T, Jacob K, Thomas J, Przetocki V, Luberice K, Sucandy I. Cost Analysis of Pancreaticoduodenectomy at a High-Volume Robotic Hepatopancreaticobiliary Surgery Program. J Am Coll Surg. 2021 Apr;232(4):461-469. doi: 10.1016/j.jamcollsurg.2020.12.062. Epub 2021 Feb 10. PMID 33581292
- [Result] Belfiori G, Crippa S, Francesca A, Pagnanelli M, Tamburrino D, Gasparini G, Partelli S, Andreasi V, Rubini C, Zamboni G, Falconi M. Long-Term Survivors after Upfront Resection for Pancreatic Ductal Adenocarcinoma: An Actual 5-Year Analysis of Disease-Specific and Post-Recurrence Survival. Ann Surg Oncol. 2021 Dec;28(13):8249-8260. doi: 10.1245/s10434-021-10401-7. Epub 2021 Jul 13. PMID 34258720
- [Result] Sucandy I, Shapera E, Syblis CC, Crespo K, Przetocki VA, Ross SB, Rosemurgy AS. Propensity score matched comparison of robotic and open major hepatectomy for malignant liver tumors. Surg Endosc. 2022 Sep;36(9):6724-6732. doi: 10.1007/s00464-021-08948-3. Epub 2022 Jan 3. PMID 34981238
- [Result] Aghayan DL, Kazaryan AM, Dagenborg VJ, Rosok BI, Fagerland MW, Waaler Bjornelv GM, Kristiansen R, Flatmark K, Fretland AA, Edwin B; OSLO-COMET Survival Study Collaborators. Long-Term Oncologic Outcomes After Laparoscopic Versus Open Resection for Colorectal Liver Metastases : A Randomized Trial. Ann Intern Med. 2021 Feb;174(2):175-182. doi: 10.7326/M20-4011. Epub 2020 Nov 17. PMID 33197213
- [Result] Fretland AA, Dagenborg VJ, Bjornelv GMW, Kazaryan AM, Kristiansen R, Fagerland MW, Hausken J, Tonnessen TI, Abildgaard A, Barkhatov L, Yaqub S, Rosok BI, Bjornbeth BA, Andersen MH, Flatmark K, Aas E, Edwin B. Laparoscopic Versus Open Resection for Colorectal Liver Metastases: The OSLO-COMET Randomized Controlled Trial. Ann Surg. 2018 Feb;267(2):199-207. doi: 10.1097/SLA.0000000000002353. PMID 28657937
- [Result] Shapera E, Sucandy I, Syblis C, Crespo K, Ja'Karri T, Ross S, Rosemurgy A. Cost analysis of robotic versus open hepatectomy: Is the robotic platform more expensive? J Robot Surg. 2022 Dec;16(6):1409-1417. doi: 10.1007/s11701-022-01375-z. Epub 2022 Feb 13. PMID 35152343
- [Result] Wecowski J, Ross SB, Jadick MF, Justice A, Sucandy I, Rosemurgy AS. THE Big Deal: An Institution's Experience with Robotic Transhiatal Esophagectomy. Am Surg. 2019 Sep 1;85(9):1061-1065. PMID 31638525
- [Result] van den Berg JW, Luketich JD, Cheong E. Oesophagectomy: The expanding role of minimally invasive surgery in oesophageal cancer. Best Pract Res Clin Gastroenterol. 2018 Oct-Dec;36-37:75-80. doi: 10.1016/j.bpg.2018.11.001. Epub 2018 Nov 21. PMID 30551859
- [Result] Giulianotti PC, Coratti A, Angelini M, Sbrana F, Cecconi S, Balestracci T, Caravaglios G. Robotics in general surgery: personal experience in a large community hospital. Arch Surg. 2003 Jul;138(7):777-84. doi: 10.1001/archsurg.138.7.777. PMID 12860761
- [Result] Sucandy I, Jacoby H, Crespo K, Syblis C, App S, Ignatius J, Ross S, Rosemurgy A. A Single Institution's Experience With Robotic Minor and Major Hepatectomy. Am Surg. 2023 May;89(5):1387-1391. doi: 10.1177/00031348211047500. Epub 2021 Nov 19. PMID 34798777
- [Result] Rosemurgy AS, Luberice K, Krill E, Castro M, Espineira GR, Sucandy I, Ross S. 100 Robotic Distal Pancreatectomies: The Future at Hand. Am Surg. 2020 Aug;86(8):958-964. doi: 10.1177/0003134820942181. Epub 2020 Aug 11. PMID 32779475
- [Result] Qu L, Zhiming Z, Xianglong T, Yuanxing G, Yong X, Rong L, Yee LW. Short- and mid-term outcomes of robotic versus laparoscopic distal pancreatosplenectomy for pancreatic ductal adenocarcinoma: A retrospective propensity score-matched study. Int J Surg. 2018 Jul;55:81-86. doi: 10.1016/j.ijsu.2018.05.024. Epub 2018 May 23. PMID 29802919